CLINICAL TRIAL: NCT01927237
Title: The Pulmonary Vascular Consequences of Divergent Strategies for Low Tidal Volume Ventilation: Hypercapnia or High Respiratory Rate?
Brief Title: Pulmonary Vascular Effects of Respiratory Rate & Carbon Dioxide
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Talmor, Edward Lowenstein Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2013P000222
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2014-08

CONDITIONS: Low Tidal Volume Ventilation; Acute Respiratory Distress Syndrome
Keywords: pulmonary artery pressure; ARDS; alveolar hypoventilation; hypercapnic acidosis; permissive hypercapnia; myocardial strain
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoventilation; Acidosis, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLR-first (Experimental): Patients in this arm will have the "hypercapnia with low respiratory rate" (HLR) strategy first. Once hypercapnia is achieved via inspired carbon dioxide, no additional changes will be made to the ventilator. Once steady-state is achieved, physiological measurements will be taken. The patient will be returned to baseline settings for a 15-minute "rest period" before starting the EHR strategy per the cross-over design.
  Interventions: Other: HLR; Other: EHR
- EHR-first (Experimental): Patients in this arm will have the "eucapnia with high respiratory rate" (EHR) strategy first. Once hypercapnia is achieved via inspired carbon dioxide, respiratory rate will be increased until PetCO2 returns to baseline or up to 35 breaths per minute, as limited by the National Heart Lung and Blood Institute (NHLBI) ARDS Network protocol. fraction of inspired oxygen inspired oxygen fraction and set tidal volume will be maintained. Once steady-state is achieved, physiological measurements will be taken. The patient will be returned to baseline settings for a 15-minute "rest period" before starting the HLR strategy per the cross-over design.
  Interventions: Other: HLR; Other: EHR

INTERVENTIONS:
Other: HLR
  Other Names: hypercapnia with low respiratory rate
Other: EHR
  Other Names: eucapnia with high respiratory rate

SUMMARY:
The purpose of this protocol is to perform serial physiological measurements and blood testing on mechanically ventilated patients comparing conditions of eucapnia and hypercapnia in the same patient. We will be testing two hypotheses: (1) while administering inspired carbon dioxide (CO2), eucapnia achieved by high respiratory rate (EHR) significantly decreases pulmonary artery pressures compared to hypercapnia with a lower respiratory rate (HLR), and (2) that EHR decreases myocardial strain compared to HLR.

DETAILED DESCRIPTION:
The purpose of this protocol is to perform serial physiological measurements and blood testing on mechanically ventilated patients comparing conditions of eucapnia (maintaining alveolar ventilation to target carbon dioxide partial pressure (pCO2) 35-40 mm Hg) and hypercapnia (providing inspired CO2 to target pCO2 55-60 mm Hg) in the same patient. This prospective clinical study will enroll consenting adult patients scheduled for elective cardiac surgery and who require postoperative mechanical ventilation, pulmonary artery (Swan-Ganz) catheter monitoring, and arterial catheterization as part of routine standard care during the immediate postoperative period. The study will perform measurements using available ventilator monitors, ventilator in-line pneumotachograph and capnograph, measurements from the indwelling pulmonary artery catheter, transesophageal echocardiography, and other measurements available as part of routine care. The entire experimental protocol will be performed in one day over 2-4 hours, and the protocol will not interfere with routine postoperative care, nor prolong the need for mechanical ventilation, pulmonary artery catheterization, arterial catheterization, or intensive care unit length of stay.

Ventilation with low tidal volumes has been shown definitively to improve mortality from acute respiratory distress syndrome (ARDS)1 and may provide benefit even in patients without ARDS.2 During low tidal volume ventilation, practice varies on whether to allow some degree of alveolar hypoventilation with incidental hypercapnic acidosis (termed "permissive hypercapnia"),3 or to increase respiratory rate to maintain alveolar ventilation and target eucapnia, often requiring respiratory rates > 30/min.4 The physiological consequences of these divergent strategies remain to be fully elucidated. We propose the following study to distinguish the effects of a eucapnic high respiratory rate (EHR) strategy from a hypercapnic low respiratory rate (HLR) strategy on pulmonary hemodynamics during low tidal volume ventilation.

Specific Aim: To test the hypothesis that, while administering inspired CO2, eucapnia achieved by high respiratory rate (EHR) significantly decreases pulmonary artery pressures compared to hypercapnia with a lower respiratory rate (HLR).

Specific Aim: To test the hypothesis that EHR decreases myocardial strain compared to HLR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Able to consent pre-operatively prior to scheduled cardiac surgery.
* Intubation on mechanical ventilation post-operatively.
* Presence of a pulmonary artery catheter and/or central venous catheter as part of usual care post-operatively.
* Presence of a radial, brachial, or femoral arterial catheter as part of usual care post-operatively.

Exclusion Criteria:

* Significant intra-operative or immediate post-operative complications, such as uncontrolled bleeding or persistent hemodynamic instability.
* Intra-cardiac or intrapulmonary shunt.
* Persistent post-operative moderate or severe hypoxemia, defined as PaO2/FiO2 < 200 mmHg.
* Moderate or severe lung disease, including moderate or severe chronic obstructive pulmonary disease (COPD) or asthma.
* Recently treated for bleeding varices, stricture, or hematemesis, esophageal trauma, recent esophageal surgery, or other contraindication to transesophageal echocardiography.
* Severe coagulopathy (platelet count < 10,000 or international normalized ratio [INR] > 4).
* History of lung, heart, or liver transplant.
* Elevated intracranial pressure or conditions where hypercapnia-induced elevations in intracranial pressure should be avoided, including:

  * Intracranial hemorrhage
  * Cerebral contusion
  * Cerebral edema
  * Mass effect (midline shift on head CT)
  * Flat EEG for > 2 hours
* Evidence of active air leak from the lung, such as broncho-pleural fistula or ongoing air leak from an existing chest tube.
* Treating physician refusal.
* Inability to obtain informed consent directly from the subject prior to surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
mean pulmonary artery pressure (mPAP) | 4 hours
  Pulmonary artery pressure will be measured directly by transducing the pulmonary artery catheter, and will include systolic (PASP) and diastolic (PADP) Ppa. The mean pulmonary artery pressure (mPAP) will be calculated according to the formula: mPAP = 1/3 PASP + 2/3 PADP

SECONDARY OUTCOMES:
Right ventricular systolic function | 4 hours
  Right ventricular systolic function will be assessed using strain echocardiography or peak tricuspid annular systolic velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra A. Low-tidal-volume ventilation in the acute respiratory distress syndrome. N Engl J Med. 2007 Sep 13;357(11):1113-20. doi: 10.1056/NEJMct074213. PMID 17855672
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162